# **Informed Consent Form**

Document data: Sep 1,2020

It is our aim to improve the quality of life in patients with tracheostomy with the respect due to individual rights in accordance with the internationally accepted ethical rules, ensuring you that all the research to be carried out will be under the supervision of an Ethical Committee, that will ensure the observance of the mentioned regulations. For the above reasons we request your voluntary collaboration.

### Purpose of the study

This study is to determine if the new tracheostomy tie is better than the old one.

#### **Procedures**

If you agree to participate in this project, you will be randomly assigned to use traditional tracheostomy tie or new one after tracheostomy. Then you will be invited to finish a questionnaire and the skin status will be recorded.

#### 3 Benefits

This is an altruistic donation, therefore no economic compensation should be obtained by the donor. However, we expect that results obtained from its use will enable us to improve the knowledge on this kind of disorders and finally may result in useful benefits for society as a whole.

#### Physical risks

No physical risks are expected.

## Confidentiality

Both the information gathered from you and research results will be confidentially treated. Data obtained will only be published in an anonymous and aggregated way, that is to say, as percentages or numerical data without identification of the participant, never in an individualized way to prevent his/her identification.

| Name: |
|-------------------------------------------------------------|
| Surname: |
| Address: |
| Signature of participant or his/her legal representative: _ |
| Date <sup>.</sup> |